CLINICAL TRIAL: NCT03647332
Title: Use of Cooled Radiofrequency for the Treatment of Hip Pain Associated With OA of the Hip Compared to Intra-articular Steroid Injections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018Stolzenberg
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Osteo Arthritis of Hip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cooled RFA treatment (Active Comparator)
  Interventions: Procedure: Cooled RFA treatment
- Steroid injection (Active Comparator)
  Interventions: Drug: Steroid Drug

INTERVENTIONS:
Procedure: Cooled RFA treatment — cooled radiofrequency ablation
  Arms: Cooled RFA treatment
Drug: Steroid Drug — steroid injection
  Arms: Steroid injection

SUMMARY:
This will be a single-center, prospective, single-blinded randomized clinical trial to investigate the effectiveness of using cooled RFA for the treatment of OA hip pain and function in subjects treated with cooled RFA compared with standard of care intra-articular steroid injections

ELIGIBILITY:
Inclusion Criteria:

* Subjects presenting with radiographic evidence of hip OA and demonstrating hip pain for at least 30 days will be targeted. Radiographic evidence of hip OA is defined as Kellegran-Lawrence grade 2-4
* Not an operative candidate as per RI joint replacement surgeon OR
* Subjects who do not desire joint replacement surgery after consultation with RI joint replacement surgeon
* Male or non-pregnant female older than 18 years of age
* willing and able to sign the IRB-approved informed consent document.

Exclusion Criteria:

* Any steroid injection in hip within 90 days
* Local infection at injection site or active systemic infection
* Anticoagulation status with inability to discontinue medication for appropriate duration for nerve blocks and RFA given proximity to major artery. (No anticoagulation contraindications for joint injection)
* AICD with inability to utilize magnet for RFA per treating cardiologist
* Body habitus does not allow for placement of longest needles and electrodes (approximately 15cm) to successfully administer treatment
* Allergy or severe renal impairment precluding iodionated contrast or magnavist injection despite standard premedication protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pain | 24 weeks following treatment
  Visual Analog Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States